CLINICAL TRIAL: NCT03844334
Title: CLEVER: CLinical EValuation of WEB 0.017 Device in Intracranial AneuRysms
Brief Title: CLinical EValuation of WEB 0.017 Device in Intracranial AneuRysms
Acronym: CLEVER
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP EMEA 18-02
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: WEB Aneurysm Embolization System — Subjects aged ≥ 18 years, but ≤ 80 years requiring treatment for single ruptured or unruptured intracranial aneurysms.

SUMMARY:
The study is an observational, European, multi-center, prospective assessment of the clinical utility of the 0.017 WEB Aneurysm Embolization System in subjects with intracranial aneurysms deemed appropriate for endovascular treatment.

DETAILED DESCRIPTION:
All eligible subjects presenting to the participating Centers will be considered for entry into the study. Up to 160 evaluable subjects meeting the study entry criteria will be enrolled.

Subjects will be followed per Institution's standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age and ≤80 years of age
2. Subject must have an intracranial aneurysm (IA),
3. Subject must sign and date Ethics Committee approved written informed consent prior to initiation of any clinical interventional procedures or when applicable, register the patient non opposition to the study data collection
4. For ruptured aneurysm, Subject with Hunt & Hess Score ≤ III

Exclusion Criteria:

1. Subject has an IA with characteristics unsuitable for endovascular treatment
2. Subject's index IA was previously treated
3. Subject has stroke-in-evolution within the prior 30 days
4. An additional aneurysm must be treated during the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The decision to use a WEB device to treat the patient has been made before and independently of the decision to include the patient in this study
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Aneurysm occlusion | 12 months
  Angiographic (conventional Angio) occlusion based on Raymond-Roy occlusion scale The Raymond-Roy occlusion classification (RROC) is an angiographic classification scheme for grading the occlusion of endovascularly treated intracranial aneurysms.
  * class I: complete obliteration
  * class II: residual neck
  * class III: residual aneurysm
Incidence of major stroke or neurological deaths | 12months
  The proportion of subjects with death of any nonaccidental cause or any major stroke within the first 30 days after treatment or major ipsilateral stroke or death due to neurologic cause from day 31 to the 1 year after treatment

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Purpan, Toulouse
- Universitätsklinikum Knappschaftskrankenhaus, Bochum, Germany
- National Institute of Clinical Neurosciences, Budapest, Hungary

REFERENCES:
- [Derived] Spelle L, Costalat V, Caroff J, Wodarg F, Fischer S, Herbreteau D, Mohlenbruch MA, Januel AC, Papagiannaki C, Klisch J, Numminen J, Rautio R, Berlis A, Mihalea C, Chalumeau V, Downer J, Cortese J, Ikka L, Gallas S, Bester M, Liebig T, Velasco S, Grimaldi L, Byrne J, Szikora I, Pierot L, Cognard C. CLinical EValuation of WEB 17 device in intracranial aneuRysms (CLEVER): procedural, 30-day and 1-year safety results for ruptured and unruptured aneurysms. J Neurointerv Surg. 2024 Nov 22;16(12):1299-1306. doi: 10.1136/jnis-2023-020866. PMID 37914392
- See also: CLinical EValuation of WEB 17 device in intracranial aneuRysms (CLEVER): procedural, 30-day and 1-year safety results for ruptured and unruptured aneurysms — https://jnis.bmj.com/content/early/2023/11/01/jnis-2023-020866.long